CLINICAL TRIAL: NCT02552303
Title: The Treatment of Insomnia Comorbid With Sleep Disordered Breathing Using Armodafinil and/or Cognitive Behavioral Therapy for Insomnia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Teva Pharmaceutical Industries, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 817800
Record Dates: First submitted 2015-09-09; First posted 2015-09-17 (Estimated); Results first posted 2017-07-31 (Actual); Last update posted 2017-07-31 (Actual); Status verified 2017-06

CONDITIONS: Sleep Apnea; Insomnia
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy; Modafinil

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (4):
- CBT for Insomnia (CBTI) + Armodafinil (Active Comparator): CBT-I with Armodafinil (active medication)
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia; Drug: Armodafinil
- CBTI + Placebo (Placebo Comparator): Cognitive Behavioral Therapy for Insomnia with Placebo medication
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia; Drug: Placebo
- Armodafinil (Active Comparator): Medication (armodafinil) only, without CBTI.
  Interventions: Drug: Armodafinil
- Placebo (Placebo Comparator): Placebo only, without CBTI.
  Interventions: Drug: Placebo

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Insomnia — Cognitive Behavioral Therapy for Insomnia.
  Other Names: CBT-I
  Arms: CBT for Insomnia (CBTI) + Armodafinil; CBTI + Placebo
Drug: Armodafinil — Active medication
  Other Names: NuVigil
  Arms: Armodafinil; CBT for Insomnia (CBTI) + Armodafinil
Drug: Placebo — Placebo for Nuvigil (armodafinil)
  Arms: CBTI + Placebo; Placebo

SUMMARY:
The purpose of this study is to assess the effects of Armodafinil, CBT-I, or the combination of the two on the sleep continuity of persons suffering from sleep disordered breathing and their adherence to CBT-I and Continuous Positive Airway Pressure (CPAP). Adults diagnosed with obstructive sleep apnea and who meet additional research and diagnostic criteria for insomnia will be recruited. Participants will submit daily sleep diaries and supplemental questionnaires as measures of study progress.

DETAILED DESCRIPTION:
Rationale:

Insomnia and sleep disordered breathing are the most common sleep disorders and they tend to be highly comorbid. When they co-occur, not only is there an increase in cumulative morbidity, but it is likely that these two diseases interact to: promote overall greater illness severity; reduce treatment adherence; and diminish treatment efficacy. The results from the proposed project will provide valuable information on how co-treatment for these two disorders can promote improved sleep quantity, enhanced sleep quality, better compliance with Positive Airway Pressure (PAP) therapy, and better daytime functioning.

Background:

There is now substantial evidence that Cognitive Behavioral Therapy for Insomnia (CBT-I) is efficacious for Primary Insomnia (PI), that it is as potent as sedative hypnotic treatment, and better sustained over time. Further, there is now increasing evidence that CBT-I can be applied to insomnias that are co-morbid with medical and psychiatric disorders, and with equal efficacy. The evidence for an expanded indication, to date, has been for insomnia comorbid with depression, chronic pain, and cancer. Interestingly, there are very few studies on the efficacy of CBT-I in insomnia comorbid with other intrinsic sleep disorders, including in patients with Sleep Disordered Breathing (SDB). This is surprising given that insomnia frequently occurs comorbidly with SDB. It is estimated that 40-60% of patients with SDB also suffer from insomnia. The lack of data regarding the applicability of CBT-I to insomnia co-morbid with SDB is likely due to the concern that CBT-I will be difficult to tolerate in patients with insomnia co-morbid with SDB given the treatment's tendency to produce acute increases in fatigue, sleepiness, and transient reductions in attention and performance. Accordingly, the investigators of this study propose to conduct a randomized, controlled trial on the effects of Armodafinil alone and in combination with CBT-I in patients with Insomnia comorbid with SDB.

Note: The choice to evaluate Armodafinil as both a monotherapy and an adjuvant therapy to CBT-I for insomnia has a firm conceptual basis and is supported by preliminary data from our group. The choice to evaluate Armodafinil in patients with insomnia co-morbid with SDB is further supported by the existing indication for sleepiness in patients with SDB.

ELIGIBILITY:
Inclusion Criteria:

* eligible subjects must have begun their CPAP treatment within the last 3 months
* current ESS (Sleepiness) Scores between 5-19
* no history of upper airway surgery (e.g. UPPP)
* able to understand written and spoken English
* able to swallow medication
* preferred sleep phase between 9:00 pm and 9:00 am
* willing to discontinue any sleep medications/over-the-counters(OTCs)/Herbals for insomnia for the 11-week study period.
* female participants must not be pregnant or breastfeeding and must agree to use two forms of birth control during the study period, as Armodafinil may interfere with hormonal birth control.
* all participants will be asked to postpone any additional or alternate treatments for their Obstructive Sleep Apnea (OSA) until after the completion of their participation in this research study.
* for other elective procedures, prospective participants are recommended to either postpone the procedure until after completion of their participation in this study, or alternatively to start the study after completion of the elective procedure.

Exclusion Criteria:

* CPAP usage exceeding three months prior to pre-screening
* suicide attempts within the last five years
* unstable medical or psychiatric illness
* cardiac abnormalities, liver, or kidney diseases
* sleep disorders other than insomnia or SDB
* evidence of active illicit substance use or fitting criteria for alcohol abuse or dependence
* use of central nervous system (CNS) active medications, antidepressants and hypnotics prescribed as sleep-aids (these medications are permitted if prescribed for mediation of symptoms other than sleep and the patient has been on a stable dosage for a minimum of one month, with no anticipation of altering their dosage during the study period.)
* inadequate language comprehension
* pregnant or breastfeeding

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2014-04; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael L Perlis, PhD, Principal Investigator — University of Pennsylvania

RESULTS

PARTICIPANT FLOW:
Period: Allocation
Arm/Group | CBT for Insomnia (CBTI) + Armodafinil | CBTI + Placebo | Armodafinil | Placebo
Started | 10 | 10 | 8 | 11
Completed | 7 | 8 | 7 | 10
Not Completed | 3 | 2 | 1 | 1
Not completed — Withdrawal by Subject | 2 | 1 | 1 | 1
Not completed — ineligible | 1 | 1 | 0 | 0
Period: Follow-Up
Arm/Group | CBT for Insomnia (CBTI) + Armodafinil | CBTI + Placebo | Armodafinil | Placebo
Started | 7 | 8 | 7 | 10
Completed | 7 | 6 | 6 | 10
Not Completed | 0 | 2 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0
Not completed — ineligible | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CBT for Insomnia (CBTI) + Armodafinil | CBTI + Placebo | Armodafinil | Placebo | Total
Number analyzed (Participants) | 10 | 10 | 8 | 11 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.2 (9.0) | 45.0 (9.8) | 48.4 (12.4) | 51.9 (7.1) | 48.2 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 5 | 7 | 24
  Male | 3 | 5 | 3 | 4 | 15
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 8 | 11 | 39

OUTCOME MEASURES:

1. Primary Outcome: The Change in Sleep Continuity From Baseline to Follow-up, as Measured by the Insomnia Severity Index (ISI).
Description: This outcome measure is based on changes in sleep continuity, as assessed by the Insomnia Severity Index (ISI), which is administered once at baseline and once at follow-up. The ISI (Morin, 1993) was used to assess perceived sleep difficulties or current insomnia symptom severity (i.e., past two weeks). The ISI is a 7-item, self-report instrument with good reliability and validity, and positively correlated with clinician-rated insomnia diagnoses (Bastien, Vallières, & Morin, 2001). Total scores on the full 7-item scale range from 0 - 28 with higher values representing greater sleep continuity disturbance or insomnia severity.
  The four different treatment groups will be compared for differences.
Time Frame: ISI is measured once at baseline and once at follow-up (8-10 weeks apart)
Measure: Mean (Standard Deviation); unit: units on a scale (ISI)
Arm/Group | CBT for Insomnia (CBTI) + Armodafinil | CBTI + Placebo | Armodafinil | Placebo
Number analyzed (Participants) | 7 | 6 | 6 | 10
units on a scale (ISI) | 13.0 (2.1) | 17.9 (0.2) | 7.7 (0.5) | 6 (1.8)

2. Secondary Outcome: Number of Subjects Who Dropped Out
Description: Drop-out rates will be calculated by the number of protocol weeks the subject completed before withdrawing from the study. Drop out rates for subjects taking active v. placebo study medication were compared.
  Withdrawal indicates subjects who were either lost-to-follow-up (LTFU), chose to withdraw (self-withdrawn), were withdrawn by the study's PI (withdrawn by the investigator).
Time Frame: up to 8 weeks of active study
Measure: Count of Participants; unit: Participants
Arm/Group | CBT for Insomnia (CBTI) + Armodafinil | CBTI + Placebo | Armodafinil | Placebo
Number analyzed (Participants) | 10 | 10 | 8 | 11
Participants | 3 | 4 | 2 | 1

ADVERSE EVENTS:
Arm/Group | CBT for Insomnia (CBTI) + Armodafinil | CBTI + Placebo | Armodafinil | Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/8 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/8 | 0/11
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/8 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No